CLINICAL TRIAL: NCT01933919
Title: A Phase 3 Study of SME3110 (Fluvoxamine Maleate) in Pediatric/Adolescent Subjects With Obsessive Compulsive Disorder
Brief Title: A Phase 3 Study of Fluvoxamine (SME3110) in Pediatric/Adolescent Patients With Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M13-970
Record Dates: First submitted 2013-08-29; First posted 2013-09-02 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-06

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Adolescent Subjects; Pediatric Subjects
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Fluvoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): In the double-blind placebo-controlled phase participants received one placebo tablet a day in week 1, then one placebo tablet twice a day (BID) in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by one tablet/day/week up to a maximum of three tablets twice a day. From weeks 7 to 10 participants received the same dose that was given during week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to two tablets/day each week.
  In the open-label long-term phase participants received 25 mg fluvoxamine once a day for the first week, 25 mg BID in week 2 followed by a flexible dose period from weeks 3 to 52 where the dose could be escalated by one tablet/day/week up to a maximum of 150 mg/day (three tablets BID). At the end of the 52-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to 50 mg/day each week.
  Interventions: Drug: Fluvoxamine maleate; Drug: Placebo
- Fluvoxamine (Experimental): In the double-blind placebo-controlled phase participants received 25 mg fluvoxamine once a day in week 1, 25 mg twice a day (BID) in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by 25 mg/day/week up to a maximum of 150 mg (three tablets BID). From weeks 7 to 10 participants received the same dose that was given during week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose of decreased by up to 50 mg/day each week.
  In the open-label long-term phase participants received 25 mg fluvoxamine once a day for the first week, 25 mg BID in week 2 followed by a flexible dose period from weeks 3 to 52 where the dose could be escalated by 25 mg/day/week up to a maximum of 150 mg/day (three tablets BID). At the end of the 52-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to 50 mg/day each week.
  Interventions: Drug: Fluvoxamine maleate

INTERVENTIONS:
Drug: Fluvoxamine maleate — Film-coated tablet containing 25 mg of fluvoxamine maleate
  Other Names: SME3110; Luvox; Depromel
Drug: Placebo — Placebo tablet matching to fluvoxamine maleate
  Arms: placebo

SUMMARY:
The objective of the first phase of this study is to evaluate the efficacy of fluvoxamine compared to placebo on change in total score of Japanese version of the Children's Yale-Brown Obsessive Compulsive Scale (JCY-BOCS) 10-item from baseline to the last observation visit (10 weeks) in pediatric/adolescent participants with obsessive compulsive disorder (OCD).

The objective of the second phase of the study is to evaluate the long-term safety and efficacy of fluvoxamine in pediatric/adolescent patients with OCD.

DETAILED DESCRIPTION:
The first phase will be conducted in a randomized, placebo-controlled, double-blind manner to evaluate the efficacy of fluvoxamine on change from baseline to the last observation visit in the JCY-BOCS 10-item total score. Eligible patients will be allocated to the fluvoxamine group or placebo group in a 1:1 ratio using the experience of fluvoxamine treatment and age as stratification factors (dynamic allocation). The first phase consists of a screening period of 1-2 weeks, a forced titration dose period of 2 weeks, a dose adjustment period of 4 weeks, a maintained dose period of 4 weeks, and a tapering dose period of 0-4 weeks.

The 2nd phase will be conducted in an open-label manner in participants who completed the first phase to evaluate the long-term safety of fluvoxamine. The 2nd phase consists of 3 periods; a forced titration dose period of 2 weeks, a flexible dose period of 50 weeks, and a tapering dose period of 0-4 weeks. After the last dose of study drug (including tapering dose period) or the early termination visit, participants will be followed for up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has at least 16 points on Japanese version of the Children's Yale-Brown Obsessive Compulsive Scale 10-item total score and at least 5 points in Obsession sub-total score and in Compulsion sub-total score respectively at the Screening period and Baseline.
2. Subject showed less than 25% reduction in Japanese version of the Children's Yale-Brown Obsessive Compulsive Scale 10-item total score at Baseline compared to the score at the Screening period (Total score at Baseline ≥ Total score at Screening х 0.75).
3. Subject has obsessive compulsive disorder symptoms at least for 2 months at informed consent.
4. Body weight: ≥ standard weight - 2 standard deviation based on the standard weight for each age in the School Health Statistical Survey 2001.
5. Subjects with parent or legal guardian who have received explanation about the purpose, procedure and meaning of the study sufficiently and is willing to give written informed consent for the subject. (if possible, written informed assent will be obtained from the subject).

Exclusion Criteria:

1. Subject has only trichotillomania (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 312.39) or nail-biting as his/her compulsive symptoms.
2. Subject has Tourette's disorder (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 307.23). However, the simple motor tic is not excluded.
3. Subject is diagnosed with the following psychiatric disorders.

   * Schizophrenia (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 295.xx) and other psychotic disorders (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 295.40 [schizophreniform disorder], 295.70 [schizoaffective disorder], 297.1 [delusional disorder], 298.8 [brief psychotic disorder], 297.3 [shared psychotic disorder], 293.xx [psychotic disorder due to… {indicate the general medical condition}], substance induced psychotic disorder, 298.9 [psychotic disorder not otherwise specified]).
   * Depressive disorders Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 296.xx [major depressive disorder], 296.2x [single episode], 296.3x [recurrent], 300.4 [dysthymic disorder], 311 [depressive disorder not otherwise specified]).
   * Bipolar disorders (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 296.xx [bipolar I disorder], 296.0x [single manic episode], 296.40 [most recent episode hypomanic], 296.4x [most recent episode manic], 296.6x [most recent episode mixed], 296.5x [most recent episode depressed], 296.7 [most recent episode unspecified], 296.89 [bipolar II disorder], 301.13 [cyclothymic disorder], 296.80 [bipolar disorder not otherwise specified]).
   * Mental retardation (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 317 [mild mental retardation], 318.0 [moderate mental retardation], 318.1 [severe mental retardation], 318.2 [profound mental retardation], 319 [mental retardation, severity unspecified]).
   * Eating disorders (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 307.1 [anorexia nervosa], 307.51 [bulimia nervosa], 307.50 [eating disorder not otherwise specified]).
   * Attention-deficit/hyperactivity disorder (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 314.xx) and attention deficit/hyperactivity disorder not otherwise specified (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 314.9).
   * Obsessive compulsive personality disorder (Diagnostic and Statistical manual of Mental Disorders Forth Edition Text Revision: 301.4).
   * Other patients with clinical neurological disorder.
4. Subject who diagnose Major Depressive Disorder by The Mini-International Neuropsychiatric Interview for Children and Adolescents (A) at the Screening period.
5. Subject has been treated with fluvoxamine within 2 months prior to informed consent. Except for the patient whose fluvoxamine dose is not fixed and the administration period of fluvoxamine is within 6 weeks.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08-14 (Actual); Primary Completion 2015-06-18 (Actual); Study Completion 2016-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susumu Matsuki, BS, Study Director — AbbVie

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 34 clinical sites in Japan.
Pre-assignment Details: Eligible participants were randomized to placebo or fluvoxamine in a 1:1 ratio. Randomization was stratified by prior fluvoxamine treatment and age (6-11 years or 12-18 years).
Groups:
- Fluvoxamine: In the double-blind placebo-controlled phase participants received 25 mg fluvoxamine once a day in week 1, 25 mg twice a day (BID) in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by 25 mg/day/week up to a maximum of 150 mg (three tablets BID). From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose of decreased by up to 50 mg/day each week.
  In the open-label long-term phase participants received 25 mg fluvoxamine once a day for the first week, 25 mg BID in week 2 followed by a flexible dose period from weeks 3 to 52 where the dose could be escalated by 25 mg/day/week up to a maximum dose of 150 mg/day (three tablets BID). At the end of the 52-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to 50 mg/day each week.
- Placebo: In the double-blind placebo-controlled phase participants received one placebo tablet a day in week 1, then one placebo tablet BID in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by one tablet/day/week up to a maximum dose of three tablets BID. From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to two tablets/day each week.
  In the open-label long-term phase participants received 25 mg fluvoxamine once a day for the first week, 25 mg BID in week 2 followed by a flexible dose period from weeks 3 to 52 where the dose could be escalated by one tablet/day/week up to a maximum of 150 mg/day (three tablets BID). At the end of the 52-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to 50 mg/day each week.
Period: Double-blind Placebo-controlled Phase
Arm/Group | Fluvoxamine | Placebo
Started | 19 | 19
Received Study Drug | 19 | 19
Completed | 19 | 15
Not Completed | 0 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Period: Open-label Long-term Phase
Arm/Group | Fluvoxamine | Placebo
Started | 19 | 15
Completed | 12 | 9
Not Completed | 7 | 6
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set for the 1st phase (FAS1) included participants who received at least one dose of study drug and had a baseline and at least one post-baseline measurement for efficacy after week 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluvoxamine | Placebo | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (2.83) | 13.3 (2.72) | 13.5 (2.74)
Age, Customized [Count of Participants; unit: Participants]
  6-11 years | 4 | 4 | 8
  12-18 years | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 9 | 11 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 19 | 18 | 37
Prior Treatment with Fluvoxamine [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 19 | 17 | 36
Japanese version of the Children's Yale-Brown Obsessive Total Score [Mean (Standard Deviation); unit: units on a scale] — The Japanese version of the Children's Yale-Brown Obsessive Compulsive Scale (JCY-BOCS) is a 10-item questionnaire assessing the severity of OCD in the past 7 days. Severity of compulsions and obsessions are rated on a scale from 0 (none) to 4 (extreme). The total score is calculated by summing the 10 individual scores and ranges from 0 to 40, where higher scores indicate more extreme symptoms.
  units on a scale | 25.4 (5.92) | 27.1 (5.48) | 26.2 (5.69)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Japanese Children's Yale-Brown Obsessive Compulsive Scale 10-item Total Score at the End of Treatment in the First Phase
Description: The Japanese version of the Children's Yale-Brown Obsessive Compulsive Scale (JCY-BOCS) is a 10-item questionnaire assessing the severity of obsessive compulsive disorder (OCD) in the past 7 days. Severity of compulsions and obsessions are rated on a scale from 0 (none) to 4 (extreme). The total score is calculated by summing the 10 individual scores and ranges from 0 to 40, where higher scores indicate more extreme symptoms.
Time Frame: Baseline and week 10
Population: Full analysis set for the 1st phase; last observation carried forward imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fluvoxamine: In the double-blind placebo-controlled phase participants received 25 mg fluvoxamine once a day in week 1, 25 mg twice a day (BID) in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by 25 mg/day/week up to a maximum of 150 mg (three tablets BID). From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose of decreased by up to 50 mg/day each week.
- Placebo: In the double-blind placebo-controlled phase participants received one placebo tablet a day in week 1, then one placebo tablet BID in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by one tablet/day/week up to a maximum dose of three tablets BID. From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to two tablets/day each week.
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale | -10.5 (5.25) | -6.6 (7.52)
Statistical Analysis 1: Comparison: Fluvoxamine vs Placebo; Test type: Superiority; p = 0.044, ANCOVA; ANCOVA with baseline JCY-BOCS (10-item) total score and age as covariates and treatment as fixed effect; LS Mean Difference (Fluvoxamine-Placebo) = -4.3, 95% CI 2-sided [-8.5 to -0.1], Standard Error of Mean 2.07 — The model included the fixed effects of treatment, with baseline JCY-BOCS (10-item) total score and age as covariates

2. Secondary Outcome: Mean Change From Baseline in the JCY-BOCS 10-item Total Score at the End of Treatment in the First Phase Stratified by Age
Description: The Japanese version of the Children's Yale-Brown Obsessive Compulsive Scale (JCY-BOCS) is a 10-item questionnaire assessing the severity of OCD in the past 7 days. Severity of compulsions and obsessions are rated on a scale from 0 (none) to 4 (extreme). The total score is calculated by summing the 10 individual scores and ranges from 0 to 40, where higher scores indicate more extreme symptoms.
Time Frame: Baseline and week 10
Population: Full analysis set for the first phase; last observation carried forward imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fluvoxamine - Ages 6-11: In the double-blind placebo-controlled phase participants aged 6 to 11 years received 25 mg fluvoxamine once a day in week 1, 25 mg twice a day (BID) in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by 25 mg/day/week up to a maximum of 150 mg (three tablets BID). From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose of decreased by up to 50 mg/day each week.
- Placebo - Ages 6-11: In the double-blind placebo-controlled phase participants aged 6 to 11 years received one placebo tablet a day in week 1, then one placebo tablet BID in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by one tablet/day/week up to a maximum dose of three tablets BID. From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to two tablets/day each week.
- Fluvoxamine - Ages 12-18: In the double-blind placebo-controlled phase participants aged 12 to 18 years received 25 mg fluvoxamine once a day in week 1, 25 mg twice a day (BID) in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by 25 mg/day/week up to a maximum of 150 mg (three tablets BID). From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose of decreased by up to 50 mg/day each week.
- Placebo - Ages 12-18: In the double-blind placebo-controlled phase participants aged 12 to 18 years received one placebo tablet a day in week 1, then one placebo tablet BID in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by one tablet/day/week up to a maximum dose of three tablets BID. From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to two tablets/day each week.
Arm/Group | Fluvoxamine - Ages 6-11 | Placebo - Ages 6-11 | Fluvoxamine - Ages 12-18 | Placebo - Ages 12-18
Number analyzed (Participants) | 4 | 4 | 15 | 14
units on a scale | -12.5 (3.00) | -10.3 (11.95) | -10.0 (5.67) | -5.6 (5.97)

3. Secondary Outcome: Mean Change From Baseline in the JCY-BOCS 10-item Total Score at the End of Treatment in the First Phase Stratified by Gender
Description: as for outcome 2
Time Frame: Baseline and week 10
Population: Full analysis set for the 1st phase; last observation carried forward imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fluvoxamine - Males: In the double-blind placebo-controlled phase male participants received 25 mg fluvoxamine once a day in week 1, 25 mg twice a day (BID) in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by 25 mg/day/week up to a maximum of 150 mg (three tablets BID). From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose of decreased by up to 50 mg/day each week.
- Placebo - Males: In the double-blind placebo-controlled phase male participants received one placebo tablet a day in week 1, then one placebo tablet BID in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by one tablet/day/week up to a maximum dose of three tablets BID. From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to two tablets/day each week.
- Fluvoxamine - Females: In the double-blind placebo-controlled phase female participants received 25 mg fluvoxamine once a day in week 1, 25 mg twice a day (BID) in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by 25 mg/day/week up to a maximum of 150 mg (three tablets BID). From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose of decreased by up to 50 mg/day each week.
- Placebo - Females: In the double-blind placebo-controlled phase female participants received one placebo tablet a day in week 1, then one placebo tablet BID in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by one tablet/day/week up to a maximum dose of three tablets BID. From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to two tablets/day each week.
Arm/Group | Fluvoxamine - Males | Placebo - Males | Fluvoxamine - Females | Placebo - Females
Number analyzed (Participants) | 9 | 11 | 10 | 7
units on a scale | -11.9 (4.68) | -7.0 (8.38) | -9.3 (5.68) | -6.0 (6.51)

4. Secondary Outcome: Mean Change From Baseline in the JCY-BOCS 10-item Total Score at Each Visit During the First Phase
Description: as for outcome 2
Time Frame: Baseline and weeks 2, 4, 6, 8 and 10
Population: Full analysis set for the 1st phase; participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale
  Week 2: number analyzed (Participants) | 19 | 17
  Week 2 | -3.9 (3.49) | -1.6 (2.29)
  Week 4: number analyzed (Participants) | 19 | 17
  Week 4 | -5.1 (4.95) | -3.2 (4.48)
  Week 6: number analyzed (Participants) | 18 | 17
  Week 6 | -8.8 (6.31) | -5.6 (5.44)
  Week 8: number analyzed (Participants) | 19 | 16
  Week 8 | -8.6 (5.01) | -7.9 (8.39)
  Week 10: number analyzed (Participants) | 18 | 16
  Week 10 | -10.8 (5.29) | -7.2 (7.77)

5. Secondary Outcome: JCY-BOCS 10-item Total Score at Each Visit During the First Phase
Description: as for outcome 2
Time Frame: Baseline and weeks 2, 4, 6, 8 and 10
Population: Full analysis set for the first phase; participants with available data at each time point. Last observation carried forward imputation was used for the last post-baseline visit assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline | 26.6 (5.51) | 27.3 (5.26)
  Week 2: number analyzed (Participants) | 19 | 17
  Week 2 | 22.7 (6.72) | 25.1 (5.83)
  Week 4: number analyzed (Participants) | 19 | 17
  Week 4 | 21.5 (7.91) | 24.2 (6.89)
  Week 6: number analyzed (Participants) | 18 | 17
  Week 6 | 17.4 (7.48) | 22.1 (8.24)
  Week 8: number analyzed (Participants) | 19 | 16
  Week 8 | 17.9 (6.27) | 19.6 (10.46)
  Week 10: number analyzed (Participants) | 18 | 16
  Week 10 | 15.4 (6.48) | 20.7 (9.80)
  Last post-baseline visit | 16.1 (6.84) | 20.7 (9.21)

6. Secondary Outcome: Percentage of Participants Much Improved in Clinical Global Impression Improvement Assessment During the First Phase
Description: The investigator evaluated Clinical Global Impression (CGI) to rate participants' clinical symptomatology according to the following seven categories at each visit compared to the day of the first dose of study medication:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Worse
  7. Very much worse
  Much improved includes CGI score categories 'very much improved' and 'much improved'.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 8, and 10
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 19 | 18
percentage of participants
  Week 1 | 0.0 | 0.0
  Week 2: number analyzed (Participants) | 19 | 17
  Week 2 | 5.3 | 0.0
  Week 3 | 5.3 | 11.1
  Week 4: number analyzed (Participants) | 19 | 17
  Week 4 | 10.5 | 5.9
  Week 5: number analyzed (Participants) | 19 | 17
  Week 5 | 26.3 | 5.9
  Week 6: number analyzed (Participants) | 18 | 17
  Week 6 | 38.9 | 29.4
  Week 8: number analyzed (Participants) | 19 | 16
  Week 8 | 42.1 | 43.8
  Week 10: number analyzed (Participants) | 18 | 16
  Week 10 | 50.0 | 43.8
  Last post-baseline visit | 52.6 | 38.9

7. Secondary Outcome: Percentage of Participants With a ≥ 25% Decrease From Baseline in JCY-BOCS (10-item) Total Score at the End of Treatment in the First Phase
Description: The Japanese version of the Children's Yale-Brown Obsessive Compulsive Scale (JCY-BOCS) is a 10-item questionnaire assessing the severity of OCD in the past 7 days. Severity of compulsions and obsessions were rated on a scale from 0 (none) to 4 (extreme). The total score was calculated by summing the 10 individual scores and ranges from 0 to 40, where higher scores indicate more extreme symptoms.
Time Frame: Baseline and week 10
Population: Full analysis set for the first phase; last observation carried forward imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 19 | 18
percentage of participants | 73.7 | 44.4

8. Secondary Outcome: Percentage of Participants With a ≥ 35% Decrease From Baseline in JCY-BOCS (10-item) Total Score at the End of Treatment in the First Phase
Description: as for outcome 7
Time Frame: Baseline and week 10
Population: Full analysis set for the first phase; last observation carried forward imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 19 | 18
percentage of participants | 68.4 | 33.3

9. Secondary Outcome: Mean Change From Baseline in the JCY-BOCS 10-item Total Score at Each Visit During the Second Phase
Description: The Japanese version of the Children's Yale-Brown Obsessive Compulsive Scale (JCY-BOCS) is a 10-item questionnaire assessing the severity of OCD in the past 7 days. Severity of compulsions and obsessions are rated on a scale from 0 (none) to 4 (extreme). The total score is calculated by summing the 10 individual scores and ranges from 0 to 40, where higher scores indicate more extreme symptoms.
  Baseline for the 2nd phase was the first visit of the 2nd phase after completion of the tapering period in the first phase and prior to study drug administration in the 2nd phase.
Time Frame: Baseline of the 2nd phase and weeks 2, 8, 16, 28, 40, and 52 of the 2nd phase
Population: The full analysis set (FAS) for the 2nd phase (FAS2) included participants who received at least one dose of study drug, and had a baseline and at last one post-baseline measurement for efficacy after week 1 in the 2nd phase. Last observation carried forward imputation was used for the last post-baseline visit assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fluvoxamine/Fluvoxamine: In the open-label long-term phase participants who received fluvoxamine in the first phase then received 25 mg fluvoxamine once a day for the first week, 25 mg fluvoxamine BID in week 2 followed by a flexible dose period from weeks 3 to 52 where the dose could be escalated by 25 mg/day/week up to a maximum dose of 150 mg/day (three tablets BID). At the end of the 52-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to 50 mg/day each week.
- Placebo/Fluvoxamine: In the open-label long-term phase participants who received placebo in the first phase then received 25 mg fluvoxamine once a day for the first week, 25 mg fluvoxamine BID in week 2 followed by a flexible dose period from weeks 3 to 52 where the dose could be escalated by one tablet/day/week up to a maximum of 150 mg/day (three tablets BID). At the end of the 52-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to 50 mg/day each week.
Arm/Group | Fluvoxamine/Fluvoxamine | Placebo/Fluvoxamine
Number analyzed (Participants) | 18 | 15
units on a scale
  Baseline of 2nd phase | 14.8 (6.62) | 20.4 (9.81)
  Change from baseline at week 2 | -0.2 (3.93) | -1.1 (6.55)
  Change from baseline at week 8 | -1.2 (2.87) | -4.3 (7.54)
  Change from baseline at week 16: number analyzed (Participants) | 14 | 14
  Change from baseline at week 16 | -1.3 (2.95) | -7.1 (8.53)
  Change from baseline at week 28: number analyzed (Participants) | 14 | 12
  Change from baseline at week 28 | -0.7 (3.87) | -6.2 (6.13)
  Change from baseline at week 40: number analyzed (Participants) | 13 | 8
  Change from baseline at week 40 | -1.9 (3.97) | -5.6 (11.02)
  Change from baseline at week 52: number analyzed (Participants) | 14 | 11
  Change from baseline at week 52 | -3.1 (4.48) | -6.6 (9.15)
  Change from baseline at last post-baseline visit | -1.7 (5.48) | -8.1 (8.61)

10. Secondary Outcome: Percentage of Participants Much Improved in Clinical Global Impression Improvement Assessment During the Second Phase
Description: The investigator evaluated Clinical Global Impression (CGI) to rate participants' clinical symptomatology according to the following seven categories at each visit compared to the day of the first dose of study medication in the 2nd phase:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Worse
  7. Very much worse
  Much improved includes CGI score categories 'very much improved' and 'much improved'.
Time Frame: Baseline of the 2nd phase and weeks 1, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Full analysis set for the 2nd phase; last observation carried forward imputation was used for the last post-baseline visit assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Fluvoxamine/Fluvoxamine | Placebo/Fluvoxamine
Number analyzed (Participants) | 19 | 15
percentage of participants
  Week 1: number analyzed (Participants) | 18 | 14
  Week 1 | 22.2 | 7.1
  Week 2: number analyzed (Participants) | 18 | 15
  Week 2 | 5.6 | 20.0
  Week 3: number analyzed (Participants) | 16 | 14
  Week 3 | 12.5 | 35.7
  Week 4: number analyzed (Participants) | 18 | 15
  Week 4 | 16.7 | 33.3
  Week 5: number analyzed (Participants) | 17 | 11
  Week 5 | 23.5 | 54.5
  Week 6: number analyzed (Participants) | 18 | 15
  Week 6 | 22.2 | 46.7
  Week 8: number analyzed (Participants) | 18 | 15
  Week 8 | 33.3 | 60.0
  Week 12: number analyzed (Participants) | 17 | 15
  Week 12 | 29.4 | 53.3
  Week 16: number analyzed (Participants) | 14 | 14
  Week 16 | 35.7 | 64.3
  Week 20: number analyzed (Participants) | 14 | 14
  Week 20 | 50.0 | 64.3
  Week 24: number analyzed (Participants) | 14 | 13
  Week 24 | 42.9 | 53.8
  Week 28: number analyzed (Participants) | 14 | 12
  Week 28 | 64.3 | 58.3
  Week 32: number analyzed (Participants) | 14 | 10
  Week 32 | 57.1 | 40.0
  Week 36: number analyzed (Participants) | 14 | 11
  Week 36 | 50.0 | 27.3
  Week 40: number analyzed (Participants) | 13 | 8
  Week 40 | 61.5 | 25.0
  Week 44: number analyzed (Participants) | 14 | 11
  Week 44 | 50.0 | 45.5
  Week 48: number analyzed (Participants) | 14 | 11
  Week 48 | 50.0 | 27.3
  Week 52: number analyzed (Participants) | 14 | 11
  Week 52 | 57.1 | 36.4
  Last post-baseline visit | 42.1 | 46.7

11. Secondary Outcome: Number of Participants With Adverse Events During the First Phase
Description: An adverse event (AE) was assessed as treatment-related by the investigator if there was evidence to suggest a causal relationship between the study drug and the adverse event.
  The investigator used the following definitions to rate the severity of each adverse event:
  Mild: The adverse event was transient and easily tolerated by the participant;
  Moderate: The adverse event caused the participant discomfort and interrupted usual activities.
  Severe: The adverse event caused considerable interference with the participant's usual activities and may have been incapacitating or life-threatening.
  A serious adverse event was any event that resulted in death, was life-threatening, resulted in hospitalization or prolongation of hospitalization, congenital anomaly, persistent or significant disability/incapacity, or was an important medical event requiring medical or surgical intervention to prevent a serious outcome.
Time Frame: From the first dose of the study drug up to 30 days after the last dose of the study drug, approximately 18 weeks in the first phase.
Population: Participants who received the study drug at least once in the first phase
Measure: Number; unit: participants
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 19 | 19
participants
  Any adverse event | 13 | 15
  Treatment-related adverse event | 6 | 5
  Severe adverse event | 0 | 0
  Serious adverse events | 0 | 0
  AE leading to discontinuation of study drug | 0 | 1
  AE leading to death | 0 | 0

12. Secondary Outcome: Number of Participants With Adverse Events During the Second Phase
Description: An adverse event was assessed as treatment-related by the investigator if there was evidence to suggest a causal relationship between the study drug and the adverse event.
  The investigator used the following definitions to rate the severity of each adverse event:
  Mild: The adverse event was transient and easily tolerated by the participant;
  Moderate: The adverse event caused the participant discomfort and interrupted usual activities.
  Severe: The adverse event caused considerable interference with the participant's usual activities and may have been incapacitating or life-threatening.
  A serious adverse event was any event that resulted in death, was life-threatening, resulted in hospitalization or prolongation of hospitalization, congenital anomaly, persistent or significant disability/incapacity, or was an important medical event requiring medical or surgical intervention to prevent a serious outcome.
Time Frame: From the first dose of the study drug up to 30 days after the last dose of the study drug, approximately 60 weeks in the second phase of the study.
Population: Participants who received the study drug at least once in the second phase.
Measure: Number; unit: participants
Arm/Group | Fluvoxamine/Fluvoxamine | Placebo/Fluvoxamine
Number analyzed (Participants) | 19 | 15
participants
  Any adverse event | 15 | 15
  Treatment-related adverse event | 7 | 7
  Severe adverse event | 0 | 0
  Serious adverse event | 0 | 1
  AE leading to discontinuation of study drug | 2 | 0
  AE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug up to 30 days after the last dose of the study drug, approximately18 weeks in the first phase of the study and 60 weeks in the second phase.
Groups:
- First Phase: Fluvoxamine: In the double-blind placebo-controlled phase participants received 25 mg fluvoxamine once a day in week 1, 25 mg twice a day (BID) in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by 25 mg/day/week up to a maximum of 150 mg (three tablets BID). From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose of decreased by up to 50 mg/day each week.
- First Phase: Placebo: In the double-blind placebo-controlled phase participants received one placebo tablet a day in week 1, then one placebo tablet BID in week 2 followed by a dose adjustment period from weeks 3 to 6 where the dose could be escalated by one tablet/day/week up to a maximum dose of three tablets BID. From weeks 7 to 10 participants received the same dose that was given in week 6. At the end of the 10-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to two tablets/day each week.
- Second Phase: Fluvoxamine/Fluvoxamine: In the open-label long-term phase participants who received fluvoxamine in the first phase then received 25 mg fluvoxamine once a day for the first week, 25 mg fluvoxamine BID in week 2 followed by a flexible dose period from weeks 3 to 52 where the dose could be escalated by 25 mg/day/week up to a maximum dose of 150 mg/day (three tablets BID). At the end of the 52-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to 50 mg/day each week.
- Second Phase: Placebo/Fluvoxamine: In the open-label long-term phase participants who received placebo in the first phase then received 25 mg fluvoxamine once a day for the first week, 25 mg fluvoxamine BID in week 2 followed by a flexible dose period from weeks 3 to 52 where the dose could be escalated by one tablet/day/week up to a maximum of 150 mg/day (three tablets BID). At the end of the 52-week treatment period there was a dose-tapering period of up to 4 weeks where the dose was decreased by up to 50 mg/day each week.
Arm/Group | First Phase: Fluvoxamine | First Phase: Placebo | Second Phase: Fluvoxamine/Fluvoxamine | Second Phase: Placebo/Fluvoxamine
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 1/15
Other Adverse Events (participants affected / at risk) | 13/19 | 15/19 | 15/19 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | First Phase: Fluvoxamine (N=19) | First Phase: Placebo (N=19) | Second Phase: Fluvoxamine/Fluvoxamine (N=19) | Second Phase: Placebo/Fluvoxamine (N=15)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | First Phase: Fluvoxamine (N=19) | First Phase: Placebo (N=19) | Second Phase: Fluvoxamine/Fluvoxamine (N=19) | Second Phase: Placebo/Fluvoxamine (N=15)
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 2
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 6 | 3 | 8
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 2 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 1 | 0
Waist circumference increased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 1 | 3 | 2
Hypomania (Psychiatric disorders) | 1 | 0 | 0 | 0
Dissociative disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Self injurious behavior (Psychiatric disorders) | 1 | 1 | 1 | 0
Withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Gastroenteritis norovirus (Gastrointestinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.